CLINICAL TRIAL: NCT01333488
Title: A Phase 2, Randomized, Controlled 2x3 Trial Comparing Clinical Outcomes in Patients With Severe Traumatic Brain Injury Using Mild Hypothermia and Concurrent and Supplemental Infusion of Magnesium Sulfate.
Brief Title: Mild Hypothermia and Supplemental Magnesium Sulfate Infusion in Severe Traumatic Brain Injury (TBI) Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Greg Zorman, Chief of Neurosurgery, United States Department of Defense
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHS TBI Study
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic; Brain; Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional Therapy (No Intervention)
- Hypothermia (Experimental): Subjects will have their core body temperatures lowered to 34C.
  Interventions: Device: Arctic Sun
- Hypothermia plus supplemental magnesium sulfate infusion (Experimental)
  Interventions: Device: Arctic Sun; Drug: Magnesium Sulfate

INTERVENTIONS:
Device: Arctic Sun — Core Body Temperature will be lowered using an Arctic Sun device to 34C. Bladder probe will monitor core temperature.
  Arms: Hypothermia; Hypothermia plus supplemental magnesium sulfate infusion
Drug: Magnesium Sulfate — IVI drug levels of Magnesium Sulfate targeted to plasma levels of magnesium of 2.5-3.5 mEq/Liter.(1.25-1.75mmol/L; or 3.04 - 4.26mg/dL)for 72 hours.
  Arms: Hypothermia plus supplemental magnesium sulfate infusion

SUMMARY:
The investigators hypothesize that hypothermia (body cooling) and additional magnesium sulfate will improve the outcome of severe Traumatic Brain Injury (TBI) patients.

This is a study to compare the outcomes of patients with severe traumatic brain injury who have been allocated to one of the following three groups:

Group 1 - Conventional therapy following traumatic brain injury Group 2 - Subjects will have their core body temperature lowered to 34C Group 3 - Subjects will have their core body temperature lowered to 34C and will receive a supplemental intravenous infusion of magnesium sulfate.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females ≥ 18 years of age
2. Subjects with Traumatic Brain Injury and a post-resuscitation Glasgow Coma Score (GCS) ≤ 8
3. In-hospital and screened within 7 hours of injury.
4. Able to obtain legally effective written consent from authorized representative
5. Patients who are intubated and on mechanical ventilation
6. Admitted to ICU

Exclusion Criteria:

1. Bladder or rectal core temperature below 32C (89.6F) upon admission
2. Clinical brain death
3. Patients with open abdomens.
4. Multiple orthopedic injuries (> 2 long bone fractures)
5. Persistent hypotension (systolic blood pressure < 90mmHg)
6. Persistent hypoxia (O2 Saturation < 94%)
7. Persistent metabolic acidosis (Lactic acid > 5 mmol/L, arterial pH < 7.25)
8. Positive serum pregnancy test
9. Cardiac arrhythmia with deleterious hemodynamic effects; heart block or myocardial damage (as shown on ECG)
10. History of abnormal renal function
11. Significant Co-morbidity (i.e. CAD;COPD; severe coagulopathy)
12. Pediatric patients (< 18 years old)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Zorman, MD, Principal Investigator — Memorial Healthcare System
Locations (1):
- Memorial Regional Hospital, Hollywood, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates from 11/3/2011 to 3/10/2014 in Level one trauma center setting. Study was closed because of low accrual.
Groups:
- Conventional Therapy: Standard of Care treatment for severe traumatic brain injury.
Period: Overall Study
Arm/Group | Conventional Therapy | Hypothermia | Hypothermia Plus Supplemental Magnesium Sulfate Infusion
Started | 2 | 1 | 3
Completed | 2 | 1 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Accrual too low to analyze
Groups:
- Conventional Therapy: Standard of care therapy for severe traumatic brain injury.
- Total: Total of all reporting groups
Arm/Group | Conventional Therapy | Hypothermia | Hypothermia Plus Supplemental Magnesium Sulfate Infusion | Total
Number analyzed (Participants) | 2 | 1 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3 | 6
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 35.5 [25 to 46] | 43 [43 to 43] | 25.6 [20 to 34] | 32 [20 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 1 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: GOS (Glasgow Outcome Score)
Description: GOS=5 (Good Recovery) - Capacity to resume normal occupational and social activities, although some there may be some minor physical or mental deficits or symptoms.
  GOS=4 (Moderate Disability) - Independent and can resume almost all activities of daily living.
  GOS=3 (Severe Disability) - No longer capable of engaging in most previous personal, social or work activities. Typically are partially or totally dependent on assistance from others in daily living.
  GOS=2 ( Persistent Vegetative State ) GOS=1 (Dead)
Time Frame: Discharge from Hospital - Within 2 months from Injury
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Conventional Therapy | Hypothermia | Hypothermia Plus Supplemental Magnesium Sulfate Infusion
Number analyzed (Participants) | 2 | 1 | 3
units on a scale | 3 [1 to 5] | 3 [3 to 3] | 3 [1 to 5]

2. Secondary Outcome: GOS
Description: GOS score
Time Frame: 12 months after injury
Measure: Mean (Full Range); unit: GOS score
Arm/Group | Conventional Therapy | Hypothermia | Hypothermia Plus Supplemental Magnesium Sulfate Infusion
Number analyzed (Participants) | 2 | 1 | 3
GOS score | 5 [5 to 5] | 5 [5 to 5] | 4 [3 to 5]

3. Secondary Outcome: Vasospasm
Description: as measured by TCD (Transcranial Doppler)
Time Frame: up to 3 months
Measure: Number; unit: Percentage of participants
Arm/Group | Conventional Therapy | Hypothermia | Hypothermia Plus Supplemental Magnesium Sulfate Infusion
Number analyzed (Participants) | 2 | 1 | 3
Percentage of participants | 100 | 0 | 66.6

ADVERSE EVENTS:
Time Frame: SAEs were collected from the time of patient enrollment onto the study to end of participation. Patients were followed for 12 months.
Description: 8 SAEs in total No non-serious AEs were collected.
Arm/Group | Conventional Therapy | Hypothermia | Hypothermia Plus Supplemental Magnesium Sulfate Infusion
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1 | 2/3
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Therapy (N=2) | Hypothermia (N=1) | Hypothermia Plus Supplemental Magnesium Sulfate Infusion (N=3)
sustained sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Left urethral Stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Low accrual leading to early termination and insufficient numbers for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must obtain permission from sponsor to publish any data related to this trial.